CLINICAL TRIAL: NCT05379556
Title: LOng COvid COmorbidities: Evaluation of Andrological, Reproductive and Sexual Functions in Patients Recovered From COVID-19
Brief Title: LOng COvid COmorbidities: Andrological, Reproductive, Sexual Dysfunctions in Patients Recovered From COVID-19
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Collaborators: Azienda Sanitaria Locale Napoli 2 Nord (Other)
Responsible Party: Principal Investigator, Prof. Rosario Pivonello, Clinical Professor, Federico II University
Other Study IDs: LO-COCO-ANDRO
Record Dates: First submitted 2022-05-16; First posted 2022-05-18 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Long Covid-19
Keywords: Long Covid-19; Andrological complications; Reproductive complications; Sexual complications; Olfactory complications
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Assessment of andrological profile of LO-COCO-ANDRO male patients — Assessment of serum prolactin (PRL), luteininzing hormone (LH), follicle stimulating hormone (FSH), 17β-estradiol, testosterone. Physical examination with measurement of body weight, height, body mass index, waist and hip circumference. Andrological physical examination with evaluation of testis volume with Prader orchidometer, testicular consistency and lesions, varicocele. Scrotal ultrasound performed in longitudinal, transverse and oblique scans using a high frequency linear probe with grayscale and color-doppler; transrectal prostate ultrasound performed with transverse, longitudinal and oblique scans using an "end fire" probe; basal penile ultrasound will be performed in longitudinal and transverse scans using a high frequency linear probe with grayscale and color-doppler; dynamic penile ultrasound performed as described for basal penile ultrasound after intra-cavernous infiltration of 10 mcg of prostaglandin-E1 (PGE1).
Diagnostic Test: Assessment of reproductive function of LO-COCO-ANDRO male patients — Semen samples will be collected on site by masturbation directly into a sterile plastic container after 3-5 days of sexual abstinence. The sample will be analyzed according to World Health Organization (WHO) 2010 guidelines. Semen samples will be stored for biochemical and molecular evaluations.
Diagnostic Test: Assessment of sexual function of LO-COCO-ANDRO male patients — Validated questionnaires to assess the prevalence of male sexual disorders, namely erectile dysfunction with International Index of Erectile function 15 (IIEF-15), premature ejaculation with premature ejaculation diagnostic tool (PEDT), hypoactive sexual desire disorder with andrological structured interview on erectile dysfunction (ANDRO-SIEDY). Patients will be also interviewed to evaluate lifestyle habits.
Diagnostic Test: Assessment of olfactory function of LO-COCO-ANDRO male and female patients — Brief interview to collect patient's anamnesis relative to olfactory function, with particular reference to hypo / anosmia and hypo/ageusia onset timeline, duration and regression.
  Interview for the self-assessment of chemosensory skills and for the evaluation of quality of life in relation to olfactory dysfunction.
  Sniffin 'Sticks test for the evaluation of odor threshold (T), odor discrimination (D) and odor identification (I) (TDI score).

SUMMARY:
Considering the compelling amount of studies focused on patients in the active phase of COVID-19 disease and the scarcity of studies focused on patient cured from disease aimed at evaluating the sequelae of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection, the purpose of the study is to investigate, in patients recovered from COVID-19 disease: 1) whether SARS-CoV-2 infection has induced in male patients, a primary (testicular) and / or secondary (pituitary) damage to the hypothalamic-pituitary-testicular hormonal axis, structural and / or functional damage to the testis and penis, sexual dysfunction or fertility disorders; 2) the prevalence in male and female patients of chemosensory symptoms (olfactory dysfunction) and assess whether there is a correlation between the prevalence, severity, duration and eventual persistence of olfactory dysfunction and the severity of COVID-19 disease. Patients will be evaluated at baseline (at discharge from infectious and/or pneumology unit) and after 3- 12 months. A better definition of the prevalence and type of sequelae after recovery from COVID-19 disease could significantly improve the therapeutic management and long-term follow-up of these patients, with a relevant impact in terms of health resources and public health.

DETAILED DESCRIPTION:
The testis is among the male organs with the highest expression of angiotensin-converting enzyme 2 (ACE2), particularly in Sertoli cells, Leydig cells, spermatogonia, spermatocytes and spermatids; therefore, the possibility of SARS-CoV-2 infection spread to the testis and of a direct damage to testicular endocrine function and spermatogenesis is not a negligible aspect. In addition, the possibility of indirect testicular damage has been suggested; indeed, orchitis has been reported in patients with SARS-CoV-2, favored by the activation of a systemic inflammatory response to SARS-CoV-2 infection, and changes in gonadotropin levels that support the presence of subclinical or compensated hypogonadism associated with SARS-CoV-2 infection have been highlighted, although the possibility of effects mediated by the inflammatory state, the use of corticosteroids or stress cannot be excluded. Controversial data are available regarding the possibility that SARS-CoV-2 infection can actually spread to semen, and there is currently no evidence of a direct association between SARS-CoV-2 infection and male infertility, although an altered expression of ACE2 has been associated with non-obstructive azoospermia. The widespread expression of ACE2 by endothelial cells represents an additional susceptibility alert in relation to the male reproductive system, as well as to sexual function, in particular for the potential direct and indirect effects of SARS-CoV-2 infection on the penile vascular endothelium; indeed, multiple evidences support the presence of a multi-organ endothelial dysfunction in SARS-CoV-2 infection, connected to the direct tropism of the virus mediated by the diffuse expression of ACE-2 in endothelial cells, as well as to the systemic inflammation through the increased production of pro-inflammatory cytokines which mediate/favor the alteration of the function and permeability of the vascular endothelium. In this context, erectile dysfunction could represent a long-term complication of Covid-19; penile vascular endothelial dysfunction is indeed recognized as the dominant mechanism in the onset of vasculogenic erectile dysfunction, and preliminary studies highlight a significantly higher prevalence of erectile dysfunction in patients with Covid-19, regardless of other variables affecting erectile function, such as psychological state, age and body mass index. Anosmia/hyposmia, associated or not with ageusia, has been frequently reported as a symptom of the onset of SARS-CoV-2 infection, but it could also remain the only clinical manifestation in some paucisymptomatic patients. The incidence of anosmia in SARS-CoV-2 patients is around values between 33.9% and 68%, with a predominance in the female sex. The etiopathogenetic mechanisms underlying the onset of anosmia in these patients are yet to be fully clarified; the main mechanisms proposed include damage to olfactory sensory neurons or direct invasion of the brain via the olfactory bulb. Smell disorders affect nutrition and quality of life with important psycho-social consequences. In this scenario, it appears of primary importance to evaluate and monitor the long-term evolution of anosmia in post SARS-CoV-2 infection through an objective assessment.

The aim of the study is to investigate whether in male patients recovered from COVID-19 disease, SARS-CoV-2 infection has induced: 1) alterations of seminal parameters (oligo-, astheno-, teratozoospermia, azoospermia, necrozoospermia, leukocytospermia, hypo / hyperposia); 2) hypogonadism; 3) morpho-structural alterations of the testis evaluated by ultrasonography (testicular hypotrophy, testicular and / or epididymal inhomogeneity, testicular calcifications / microlithiasis, testicular solid lesions, hydrocele, varicocele, altered testicular and / or epididymal vascularization); 4) prostate-vesicular morpho-structural alterations assessed by ultrasonography; 5) morpho-structural and hemodynamic alterations of the penis evaluated by ultrasonography with Color and PowerDoppler performed at baseline, and in some selected cases which will be identified as pathological at baseline, also performed dynamically after intra-cavernous infiltration of prostaglandin-E1 (PGE1) (morphological alterations, nodules, alterations of the albuginea tunic, presence of fibrotic or calcified plaques, morphological and haemodynamic alterations of the cavernous arteries, anastomosis between the cavernous arteries and the dorsal artery, presence of other collateral circulation, presence and site of any occlusions); 6)male sexual dysfunctions (erectile dysfunction, premature ejaculation, hypoactive sexual desire disorder) assessed by sexological questionnaires. Moreover, the aim of the study is also to investigate whether in male and female patients recovered from COVID-19 disease, SARS-CoV-2 infection has induced an olfactory dysfunction, with evaluation of the eventual correlation between prevalence, severity, duration and possible permanence of olfactory dysfunction and the severity of the COVID-19 disease, using the Sniffin 'Sticks test for the evaluation of: odor threshold (T), odor discrimination (D) and odor identification (I) (TDI score).

Patients will be evaluated at baseline (at discharge from infectious and/or pneumology unit) and after 3- 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes recovered from SARS-CoV-2 infection (two negative nasopharyngeal swabs, negative IgM and positive anti SARS-CoV-2 IgG);
* Aged over 18 years of age;
* Ability to understand protocol procedures

Exclusion Criteria:

* Any psychological/psychiatric/other medical conditions compromising the understanding of the nature and purpose of the study, and of its possible consequences
* Uncooperative attitude of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients of both sexes recovered from SARS-CoV-2 infection
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-27 (Actual); Primary Completion 2026-01-27 (Estimated); Study Completion 2027-01-27 (Estimated)

PRIMARY OUTCOMES:
Identification of the most frequent phenotypes of Long-COVID syndrome among COVID-19 patients recently hospitalized and dismissed | Change from baseline at 3-12 months
  This pilot study will allow identifying the frequency and type of andrological, reproductive, sexual and olfactory disorders that contribute to the long covid syndrome.

SECONDARY OUTCOMES:
Number of patients with andrological dysfunctions | Change from baseline at 3-12 months
  Prevalence of andrological dysfunctions (hypogonadism, morpho-structural alterations of the testis including testicular hypotrophy, testicular and / or epididymal inhomogeneity, testicular calcifications / microlithiasis, testicular solid lesions, hydrocele, varicocele, altered testicular and / or epididymal vascularization, prostate-vesicular morpho-structural alterations, morpho-structural and hemodynamic alterations of the penis including nodules, alterations of the albuginea tunic, presence of fibrotic or calcified plaques, morphological and haemodynamic alterations of the cavernous arteries, anastomosis between the cavernous arteries and the dorsal artery, collateral circulation, occlusions).
Number of patients with reproductive dysfunctions | Change from baseline at 3-12 months
  Prevalence of male reproductive dysfunctions: alterations of seminal parameters (oligo-, astheno-, teratozoospermia, azoospermia, necrozoospermia, leukocytospermia, hypo / hyperposia).
Number of patients with sexual dysfunctions | Change from baseline at 3-12 months
  Prevalence of male sexual dysfunctions (erectile dysfunction, premature ejaculation, hypoactive sexual desire disorder).
Number of patients with olfactory dysfunctions | Change from baseline at 3-12 months
  Prevalence of olfactory dysfunctions (hypo/anosmia and hypo/ageusia) in male and female patients.

CONTACTS AND LOCATIONS:
Overall Officials: Rosario Pivonello, Prof., Principal Investigator — Federico II University
Locations (1):
- Federico II University of Naples, Naples, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cardona Maya WD, Du Plessis SS, Velilla PA. SARS-CoV-2 and the testis: similarity with other viruses and routes of infection. Reprod Biomed Online. 2020 Jun;40(6):763-764. doi: 10.1016/j.rbmo.2020.04.009. Epub 2020 Apr 17. PMID 32362571
- [Background] Chen F, Lou D. Rising Concern on Damaged Testis of COVID-19 Patients. Urology. 2020 Aug;142:42. doi: 10.1016/j.urology.2020.04.069. Epub 2020 Apr 25. No abstract available. PMID 32343996
- [Background] Corona G, Baldi E, Isidori AM, Paoli D, Pallotti F, De Santis L, Francavilla F, La Vignera S, Selice R, Caponecchia L, Pivonello R, Ferlin A, Foresta C, Jannini EA, Lenzi A, Maggi M, Lombardo F. SARS-CoV-2 infection, male fertility and sperm cryopreservation: a position statement of the Italian Society of Andrology and Sexual Medicine (SIAMS) (Societa Italiana di Andrologia e Medicina della Sessualita). J Endocrinol Invest. 2020 Aug;43(8):1153-1157. doi: 10.1007/s40618-020-01290-w. Epub 2020 May 27. PMID 32462316
- [Background] Douglas GC, O'Bryan MK, Hedger MP, Lee DK, Yarski MA, Smith AI, Lew RA. The novel angiotensin-converting enzyme (ACE) homolog, ACE2, is selectively expressed by adult Leydig cells of the testis. Endocrinology. 2004 Oct;145(10):4703-11. doi: 10.1210/en.2004-0443. Epub 2004 Jul 1. PMID 15231706
- [Background] Illiano E, Trama F, Costantini E. Could COVID-19 have an impact on male fertility? Andrologia. 2020 Jul;52(6):e13654. doi: 10.1111/and.13654. Epub 2020 May 21. PMID 32436229
- [Background] Li D, Jin M, Bao P, Zhao W, Zhang S. Clinical Characteristics and Results of Semen Tests Among Men With Coronavirus Disease 2019. JAMA Netw Open. 2020 May 1;3(5):e208292. doi: 10.1001/jamanetworkopen.2020.8292. PMID 32379329
- [Background] Liu X, Chen Y, Tang W, Zhang L, Chen W, Yan Z, Yuan P, Yang M, Kong S, Yan L, Qiao J. Single-cell transcriptome analysis of the novel coronavirus (SARS-CoV-2) associated gene ACE2 expression in normal and non-obstructive azoospermia (NOA) human male testes. Sci China Life Sci. 2020 Jul;63(7):1006-1015. doi: 10.1007/s11427-020-1705-0. Epub 2020 Apr 30. PMID 32361911
- [Background] Massarotti C, Garolla A, Maccarini E, Scaruffi P, Stigliani S, Anserini P, Foresta C. SARS-CoV-2 in the semen: Where does it come from? Andrology. 2021 Jan;9(1):39-41. doi: 10.1111/andr.12839. Epub 2020 Jul 28. PMID 32533891
- [Background] Pan F, Xiao X, Guo J, Song Y, Li H, Patel DP, Spivak AM, Alukal JP, Zhang X, Xiong C, Li PS, Hotaling JM. No evidence of severe acute respiratory syndrome-coronavirus 2 in semen of males recovering from coronavirus disease 2019. Fertil Steril. 2020 Jun;113(6):1135-1139. doi: 10.1016/j.fertnstert.2020.04.024. Epub 2020 Apr 17. PMID 32482249
- [Background] Paoli D, Pallotti F, Colangelo S, Basilico F, Mazzuti L, Turriziani O, Antonelli G, Lenzi A, Lombardo F. Study of SARS-CoV-2 in semen and urine samples of a volunteer with positive naso-pharyngeal swab. J Endocrinol Invest. 2020 Dec;43(12):1819-1822. doi: 10.1007/s40618-020-01261-1. Epub 2020 Apr 23. PMID 32329026
- [Background] Wang Z, Xu X. scRNA-seq Profiling of Human Testes Reveals the Presence of the ACE2 Receptor, A Target for SARS-CoV-2 Infection in Spermatogonia, Leydig and Sertoli Cells. Cells. 2020 Apr 9;9(4):920. doi: 10.3390/cells9040920. PMID 32283711
- [Background] Wenham C, Smith J, Morgan R; Gender and COVID-19 Working Group. COVID-19: the gendered impacts of the outbreak. Lancet. 2020 Mar 14;395(10227):846-848. doi: 10.1016/S0140-6736(20)30526-2. Epub 2020 Mar 6. No abstract available. PMID 32151325
- [Background] Xu J, Qi L, Chi X, Yang J, Wei X, Gong E, Peh S, Gu J. Orchitis: a complication of severe acute respiratory syndrome (SARS). Biol Reprod. 2006 Feb;74(2):410-6. doi: 10.1095/biolreprod.105.044776. Epub 2005 Oct 19. PMID 16237152
- [Background] Nishiga M, Wang DW, Han Y, Lewis DB, Wu JC. COVID-19 and cardiovascular disease: from basic mechanisms to clinical perspectives. Nat Rev Cardiol. 2020 Sep;17(9):543-558. doi: 10.1038/s41569-020-0413-9. Epub 2020 Jul 20. PMID 32690910
- [Background] Sansone A, Mollaioli D, Ciocca G, Limoncin E, Colonnello E, Vena W, Jannini EA. Addressing male sexual and reproductive health in the wake of COVID-19 outbreak. J Endocrinol Invest. 2021 Feb;44(2):223-231. doi: 10.1007/s40618-020-01350-1. Epub 2020 Jul 13. PMID 32661947
- [Background] Caretta N, De Rocco Ponce M, Minicuci N, Palego P, Valente U, Garolla A, Ferlin A, Foresta C. Penile doppler ultrasound predicts cardiovascular events in men with erectile dysfunction. Andrology. 2019 Jan;7(1):82-87. doi: 10.1111/andr.12561. Epub 2018 Nov 8. PMID 30407754
- [Background] Varela CG, Yeguas LAM, Rodriguez IC, Vila MDD. Penile Doppler Ultrasound for Erectile Dysfunction: Technique and Interpretation. AJR Am J Roentgenol. 2020 May;214(5):1112-1121. doi: 10.2214/AJR.19.22141. Epub 2020 Jan 28. PMID 31990215
- [Background] Sansone A, Mollaioli D, Ciocca G, Colonnello E, Limoncin E, Balercia G, Jannini EA. "Mask up to keep it up": Preliminary evidence of the association between erectile dysfunction and COVID-19. Andrology. 2021 Jul;9(4):1053-1059. doi: 10.1111/andr.13003. Epub 2021 Mar 30. PMID 33742540
- [Background] Kloner RA. Erectile dysfunction as a predictor of cardiovascular disease. Int J Impot Res. 2008 Sep-Oct;20(5):460-5. doi: 10.1038/ijir.2008.20. Epub 2008 May 15. PMID 18480824
- [Background] Corona G, Forti G, Maggi M. Why can patients with erectile dysfunction be considered lucky? The association with testosterone deficiency and metabolic syndrome. Aging Male. 2008 Dec;11(4):193-9. doi: 10.1080/13685530802468497. PMID 19172551
- [Background] Zubair AS, McAlpine LS, Gardin T, Farhadian S, Kuruvilla DE, Spudich S. Neuropathogenesis and Neurologic Manifestations of the Coronaviruses in the Age of Coronavirus Disease 2019: A Review. JAMA Neurol. 2020 Aug 1;77(8):1018-1027. doi: 10.1001/jamaneurol.2020.2065. PMID 32469387
- [Background] Hopkins C, Surda P, Kumar N. Presentation of new onset anosmia during the COVID-19 pandemic. Rhinology. 2020 Jun 1;58(3):295-298. doi: 10.4193/Rhin20.116. PMID 32277751
- [Background] Klopfenstein T, Kadiane-Oussou NJ, Toko L, Royer PY, Lepiller Q, Gendrin V, Zayet S. Features of anosmia in COVID-19. Med Mal Infect. 2020 Aug;50(5):436-439. doi: 10.1016/j.medmal.2020.04.006. Epub 2020 Apr 17. PMID 32305563
- [Background] Tong JY, Wong A, Zhu D, Fastenberg JH, Tham T. The Prevalence of Olfactory and Gustatory Dysfunction in COVID-19 Patients: A Systematic Review and Meta-analysis. Otolaryngol Head Neck Surg. 2020 Jul;163(1):3-11. doi: 10.1177/0194599820926473. Epub 2020 May 5. PMID 32369429
- [Background] Lechien JR, Chiesa-Estomba CM, De Siati DR, Horoi M, Le Bon SD, Rodriguez A, Dequanter D, Blecic S, El Afia F, Distinguin L, Chekkoury-Idrissi Y, Hans S, Delgado IL, Calvo-Henriquez C, Lavigne P, Falanga C, Barillari MR, Cammaroto G, Khalife M, Leich P, Souchay C, Rossi C, Journe F, Hsieh J, Edjlali M, Carlier R, Ris L, Lovato A, De Filippis C, Coppee F, Fakhry N, Ayad T, Saussez S. Olfactory and gustatory dysfunctions as a clinical presentation of mild-to-moderate forms of the coronavirus disease (COVID-19): a multicenter European study. Eur Arch Otorhinolaryngol. 2020 Aug;277(8):2251-2261. doi: 10.1007/s00405-020-05965-1. Epub 2020 Apr 6. PMID 32253535
- [Background] Baig AM, Khaleeq A, Ali U, Syeda H. Evidence of the COVID-19 Virus Targeting the CNS: Tissue Distribution, Host-Virus Interaction, and Proposed Neurotropic Mechanisms. ACS Chem Neurosci. 2020 Apr 1;11(7):995-998. doi: 10.1021/acschemneuro.0c00122. Epub 2020 Mar 13. PMID 32167747
- [Background] Deems DA, Doty RL, Settle RG, Moore-Gillon V, Shaman P, Mester AF, Kimmelman CP, Brightman VJ, Snow JB Jr. Smell and taste disorders, a study of 750 patients from the University of Pennsylvania Smell and Taste Center. Arch Otolaryngol Head Neck Surg. 1991 May;117(5):519-28. doi: 10.1001/archotol.1991.01870170065015. PMID 2021470
- [Background] Pence TS, Reiter ER, DiNardo LJ, Costanzo RM. Risk factors for hazardous events in olfactory-impaired patients. JAMA Otolaryngol Head Neck Surg. 2014 Oct;140(10):951-5. doi: 10.1001/jamaoto.2014.1675. PMID 25170573
- [Background] Meng X, Deng Y, Dai Z, Meng Z. COVID-19 and anosmia: A review based on up-to-date knowledge. Am J Otolaryngol. 2020 Sep-Oct;41(5):102581. doi: 10.1016/j.amjoto.2020.102581. Epub 2020 Jun 2. PMID 32563019